CLINICAL TRIAL: NCT05910203
Title: The Effect of Education Based on Health Belief Model on Smoking Perceptions and Behaviors of Visually Impaired Individuals
Brief Title: The Effect of Education Based on Health Belief Model on Smoking Behaviors of Visually Impaired Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Collaborators: Aksaray University (Other)
Responsible Party: Principal Investigator, Funda Tuncer Sahin, Lecturer, Cumhuriyet University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CumhuriyetU Health Sc
Record Dates: First submitted 2023-04-16; First posted 2023-06-18 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Smoking; Blind Eye; Health Risk Behaviors
Keywords: Visually impaired individuals; Health belief model; Nursing; Smoking
MeSH Terms: conditions — Smoking; Blindness; Health Risk Behaviors

STUDY DESIGN:
Intervention Model Description: The research was designed experimentally with "pretest-posttest control group".
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health belief model smoking cessation scale (Other): Describing the thoughts and behaviors of visually impaired individuals about quitting smoking
  Interventions: Other: The effectiveness of education
- Nicotine addiction scale (Other): Evaluation of individuals' smoking cessation status
  Interventions: Other: The effectiveness of education

INTERVENTIONS:
Other: The effectiveness of education — Training will be provided on smoking cessation.
  Other Names: Quit smoking

SUMMARY:
Health is a main human right and a need for every human being. However, due to some congenital or acquired reasons, individuals may be disabled and cannot participate in social life at the same level as their normally developing peers. The gradual increase in the world population, the advances in the treatment of chronic diseases and the prolongation of life expectancy at birth, along with the increase in economic, social and psychological problems and deterioration in environmental conditions show that the number of disabled individuals will increase in the future. Diseases caused by the use of tobacco and tobacco products rank first among preventable diseases in the world, and tobacco use is a very important public health problem. Nurses use various models developed as a guide in developing goals for lifestyle change in individuals and in interventions to achieve this. One of the studies they conduct based on the models is smoking cessation. It is believed that the studies to be carried out will strengthen the perceptions of individuals about protecting and improving their health and will guide the way in which the obstacles to smoking cessation can be perceived and resolved more easily. Based on this, it is thought that the smoking cessation study to be carried out by using HBM in visually impaired individuals will draw attention to unhealthy lifestyle behaviors and smoking addiction, which is one of these behaviors. The study was designed experimentally with "pretest-posttest control group". Before and after the planned smoking cessation training given based on HBM, the scores of Fagerström Nicotine Dependence Test and the smoking cessation scale according to HBM and hemoglobin and CO measurement values of the visually impaired individuals will be compared. Statistical package program will be used for coding, statistical analysis and evaluation of the data to be obtained from the study. T-test will be used in independent groups and t-test in dependent groups depending on the distribution features of the data in the statistical analysis. The normality distribution of the data will be evaluated by Wilk's, Kurtosis and Skewness coefficients. In the data distributed normally, non-parametric tests, Kruskal Wallis test or Mann-Whitney test will be used, and parametric tests, dependent and independent groups' t-test in two variables and ANOVA (analysis of variance) will be used in two or more variables.

DETAILED DESCRIPTION:
Health is a basic human right and need for every human being, but individuals may be disabled due to some congenital or acquired reasons. Disability is defined as a person's difficulty in adapting to social life and meeting their daily needs due to the loss of their physical, mental, spiritual, sensory and social abilities at various degrees, and therefore needing support in different areas. From a sociological point of view, a disabled individual is an individual whose accessibility is limited not because of health-related problems, but rather as a result of social pressures. In the World Health Organization (WHO) 2011 World Disability Report, it is stated that 15.6% of the population over the age of 18 worldwide is a disabled person. According to the statistics of two thousand twenty one; There are 284,366 visually impaired individuals in our country. The ratio of visually impaired individuals to the total number of disabled individuals is 10% (Statistics Bulletin of the Disabled and Elderly, December 2021). Visually impaired individuals are those who have complete or partial vision loss or impairment in one or both eyes. The inability to notice the presence or movement of an object in a certain area from the environment, the inability to notice faint shapes or letters, the inability to distinguish shapes or letters that should be visible from a distance of 6 meters, no matter what glasses are worn, means "low vision-visibility insufficiency". In other words, low vision is the state of not being able to see what a "normal" person of the same age can see, and this cannot be achieved no matter what glasses are worn. The gradual increase in the world population, the advances in the treatment of chronic diseases, the prolongation of life expectancy at birth, the increase in economic, social and psychological problems and the deterioration in environmental conditions indicate that the number of disabled individuals will increase in the future. The increase in the number of disabled individuals brings with it an increase in the problems faced by disabled individuals. Disabled individuals are placed among disadvantaged groups in society and face negative discrimination in terms of participation in social life, access to education opportunities, work and employment. Accordingly, individuals with disabilities may be poor, deprived of social security, and have difficulties in accessing and receiving health services. In the reports published recently, it is reported that the health level of individuals with disabilities is lower than the other segments of the society (United Nations, 2020).

Recent epidemiological studies indicate that low diet quality, smoking and alcohol use, and low physical activity are directly related to an increased risk of eye diseases. In addition, there are data that smoking reduces visual acuity and the perception of the brightness of colors in visually impaired individuals. Although smoking is one of the most common habits in the world, it causes deterioration of people's health with the harmful substances it contains and even causes death of individuals. Every year, many people lose their health due to smoking or exposure to cigarette smoke. In addition, physical inactivity In addition to an unhealthy diet, tobacco and tobacco products use, which is responsible for approximately 80% of the problems that cause disability such as coronary heart disease and cerebrovascular diseases, ranks first among the causes of preventable diseases. Smoking is an important public health problem that causes an increase in the burden of disease. Studies have shown that risky behaviors that negatively affect health, such as smoking, unhealthy diet, and insufficient physical activity, are more common in disabled individuals than in healthy individuals. According to the study conducted in the USA, it was concluded that 24.6% of disabled individuals are addicted to cigarettes. In addition to the lack of data on why disabled individuals start smoking, there are also studies showing that social environment and family attitudes have an effect on smoking behavior. In addition, disabled individuals who may encounter situations of not being accepted by the society may have psychological problems and may turn to cigarettes as a coping mechanism. Recent epidemiological studies indicate that low diet quality, smoking and alcohol use, and low physical activity are directly related to an increased risk of eye diseases. In addition, there are studies showing that smoking reduces visual acuity and the perception of the brightness of colors in visually impaired individuals. Programs for risky groups such as children, women and disabled individuals, who are special targets in terms of tobacco use, are becoming widespread throughout the world within the scope of combating tobacco. To ensure a comprehensive tobacco control program, continuity of community-based smoking cessation programs is required. Health professionals working in primary care, especially public health nurses, have important duties in ensuring continuity. In the programs developed, especially public health nurses are required to reach disabled people and provide counseling and guidance that disabled people need. Improving the health of individuals with disabilities and bringing them into society is possible through the education of individuals, the education of families, and the provision of health and care services to the disabled child as a whole (Çoban and Özcebe, 2019). In addition to their educational role, public health nurses have roles in providing counseling to disabled people, providing the support tools needed by disabled people, and reintegrating them into society. With the roles they fulfill while improving the health of disabled people, they can raise awareness about creating the perception of health and illness of disabled people (Emlek Sert, 2021). With the appropriate risk assessment, the public health nurse can eliminate the vulnerable-risk individuals in the society and the disabled individuals, who are one of these groups, before their health problems develop, and they can preserve their existing skills with screening and treatment practices. In addition, public health nurses should develop a relationship of trust with the individual, advocate, be a teacher and role model for the individual, and increase the capacity of individuals. In addition, they should raise awareness of disabled individuals in the society and work with vulnerable groups when necessary. Public health nurses should provide guidance on changing lifestyles (healthy lifestyle practices such as nutrition and physical activity) to improve the health of individuals with disabilities. Disabled individuals, especially visually impaired individuals, may have problems in accessing health services. Visually impaired individuals who do not have the ability to move independently and cannot go out on their own may not want to go to a health institution they have not been to before, because of the anxiety of having problems, or they may not know which institution or unit to apply for their health problems. At this point, public health nurses are required to provide the disabled individuals with the necessary counseling in the field of health in their environment. In addition, nurses should establish a relationship of trust with disabled individuals and give the message that they are available when they need it. Nurses benefit from the models developed as a guide in the interventions aimed at developing goals for lifestyle change in individuals and realizing it. One of their studies based on models is smoking cessation. Nurses benefit from multiple different behavior modification models in their interventions for smoking cessation. In addition to smoking cessation models, they can also use peer education, training on smoking addiction and the harms of smoking, and motivational interview techniques.

Studies show that nursing practices, which are made by taking the change stages of the transtheoretic model (TTM), which is used as a guide in facilitating behavior change, are one of the guiding models that can enable the individual to better understand the reasons for change and/or not change, and can facilitate behavior change. When TTM is applied considering the stages of change, it appears as one of the models that have been proven to have a positive effect on individuals' smoking cessation behavior. Another model that nurses take as a guide for smoking cessation is the Health Belief Model. The Health Belief Model (HBM) is frequently used today to explain the actions taken to protect and improve health. The model, which focuses on perceived health risks, explains screening behaviors and also explains patient behavior, patient role behaviors and the factors that facilitate the realization of health behaviors. The Health Belief Model (HBM) is frequently used in studies related to screening and early diagnosis such as breast self-examination. HBM is effectively used in the management of chronic diseases such as diabetes mellitus, in the Covid-19 vaccine and other vaccines, in protecting and promoting the health of individuals.

Although HBM is not a preferred model in studies on smoking or smoking cessation, it has recently been used to prevent negative health-related behaviors such as smoking. It is thought that the studies to be carried out will strengthen the perceptions of individuals about protecting and improving their health and will guide the way in which the obstacles in front of smoking cessation can be perceived and resolved more easily.

In the studies carried out with education and counseling for visually impaired individuals, the observation list was used during the training, and improvements were recorded in the visually impaired individuals after the training. In addition, it has been determined that the training and consultancy activities given to the visually impaired individuals on the subjects they need are beneficial for the development of the visually impaired individuals and they are more willing to solve their current problems. It has been concluded that the education given after the needs analysis of individuals makes their lives easier in their daily lives.

The purpose of this research; The purpose of this study will be to determine the effect of the planned education based on the health belief model on the smoking perception and behavior of visually impaired individuals. of the study; It is thought that it will draw attention to unhealthy lifestyle behaviors in disabled individuals and smoking addiction, which is one of these behaviors, and that the findings to be obtained from the study may guide nurses and health policies that can be developed in this direction on the effectiveness of SIM-based planned education and counseling approach, especially in gaining healthy lifestyle behaviors in visually impaired individuals. In addition, it is thought that nurses who will work with disabled individuals can be an example for reaching and approaching disabled individuals.

ELIGIBILITY:
Inclusion Criteria:

* Being visually impaired
* Be over 18 years old
* Demonstrate normal mental and cognitive development
* Smoking at least 1 cigarette in the last 30 days

Exclusion Criteria:

* Be under the age of 18
* Individuals who do not show normal development mentally and cognitively
* Non-smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of smoking cessation education based on the health belief model | 0.months- 6. months
  The data of the study; Personal Information Form prepared by the researcher will be collected using Fagerström Nicotine Dependence Test and smoking cessation scale according to the health belief model. Statistical package program will be used in coding, statistical analysis and evaluation of data. In addition to the mean, standard deviation, numbers and percentages will also be used in the evaluation of the data. At the beginning of the study, the scale and test score and hemoglobin and CO measurement values obtained in the 1st, 3rd and 6th months will be compared.
Hemoglobin measurement | 0.months- 6. months
  Hemoglobin measurement of the visually impaired individuals included in the study will be measured and their smoking status will be determined and recorded. At the beginning of the study, hemoglobin measurement values obtained in the 1st, 3rd and 6th months will be compared. Hemoglobin will be evaluated in grams per 1 deciliter.
Carbon monoxide (CO) measurement | 0.months- 6. months
  Carbon monoxide (CO) measurement of the visually impaired individuals included in the study will be measured and their smoking status will be determined and recorded. At the beginning of the study, CO measurement values obtained in the 1st, 3rd and 6th months will be compared. CO will be measured and recorded in mg/m3 or ppm.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Tuncer Şahin, Study Chair — Aksaray University
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No